CLINICAL TRIAL: NCT00003868
Title: Radiolabeled BC8 (Anti-CD45) Antibody Combined With Cyclophosphamide and Total Body Irradiation Followed by HLA-matched Related or Unrelated Stem Cell Transplantation as Treatment for Advanced Acute Myeloid Leukemia and Myelodysplastic Syndrome
Brief Title: Radiolabeled Monoclonal Antibody, Cyclophosphamide, and Total Body Irradiation Followed By Donor Stem Cell Transplantation in Treating Patients With Advanced Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1297.00; FHCRC-1297.00; NCI-H99-0028; CDR0000067032 (Registry Identifier: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2003-10-07 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Leukemia
Keywords: recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; secondary acute myeloid leukemia; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Congenital Abnormalities | interventions — Cyclophosphamide; Methotrexate; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: methotrexate
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: iodine I 131 monoclonal antibody BC8
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies can locate cancer cells and either kill them or deliver radioactive cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy work in different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Donor stem cell transplantation may be able to replace immune cells that were destroyed by radiolabeled monoclonal antibody therapy, chemotherapy and radiation therapy.

PURPOSE: Phase II trial to study the effectiveness of combining radiolabeled monoclonal antibody with cyclophosphamide and total-body irradiation followed by donor stem cell transplantation in treating patients who have advanced acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy, in terms of overall survival and disease-free survival, and toxicity of cyclophosphamide and total body irradiation in patients with acute myeloid leukemia beyond first remission receiving HLA-matched related or unrelated hematopoietic stem cell transplantation.
* Determine the maximum tolerated dose (MTD) of iodine I 131 monoclonal antibody BC8 (I131 MOAB BC8) in these patients.
* Estimate the MTD of radiation delivered by I 131 MOAB BC8 to marrow of these patients and assess the effects on growth of marrow stroma in vitro.

OUTLINE: This is radiation dose-escalation study. Patients are stratified according to available donor (related vs unrelated).

Patients receive a biodistribution dose of iodine I 131 monoclonal antibody BC8 (I131 MOAB BC8) IV, then a therapeutic dose of I131 MOAB BC8 IV 6-14 days later (day -12). Patients undergo total body irradiation twice daily on days -6 to -4. Patients receive cyclophosphamide IV on days -3 and -2. Bone marrow cells (or peripheral blood stem cells) are infused on day 0.

Patients with CNS leukemic involvement receive intrathecal methotrexate twice before the transplantation then every other week for 8 weeks beginning on day 32. These patients also receive cranial irradiation beginning on day 32.

Cohorts of 4 patients each receive escalating doses of iodine I 131 attached to a standard dose of monoclonal antibody BC8 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the radiation dose preceding that at which 2 of up to 6 patients experience graft failure.

Patients are followed at 6, 9, and 12 months, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 40 patients (20 per stratum) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Acute myeloid leukemia (AML) beyond first remission OR with primary refractory disease
  * AML that has transformed from myelodysplastic syndromes, if induction chemotherapy not recommended
* Documented CD45 expression in patients with relapsed disease

  * Not needed for patients in remission
* Circulating blast count less than 10,000/mm^3 (may be controlled with hydroxyurea or similar agent)

PATIENT CHARACTERISTICS:

Age

* 2 to 55

Performance status

* Not specified

Life expectancy

* More than 60 days

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin less than 1.5 mg/dL (unless bilirubin is determined by the gastroenterology service to be predominantly unconjugated [indirect] as the result of possible hemolysis)
* AST less than 1.5 times upper limit of normal (ULN)

Renal

* Creatinine less than 2.0 mg/dL OR less than 1.5 times ULN for age

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No major infection
* No circulating antibodies to mouse immunoglobulins
* HIV negative
* Able to tolerate diagnostic or therapeutic procedures (e.g., radiation isolation)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* No radiotherapy to maximum tolerated levels to any normal organ

Surgery

* Not specified

Ages: 2 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 1999-02; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eneida Nemecek, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States